CLINICAL TRIAL: NCT02297269
Title: The Impact of Laparoscopic Versus Open Surgeries on the Incidence of Postoperative Deep Vein Thrombosis in Patients With Gastrointestinal Malignancy ---A Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, Department of Anesthesiology and Pain Medicine, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: CYYYMZ-004
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Surgery; gastrointestinal malignancy
MeSH Terms: conditions — Venous Thrombosis | interventions — Laparoscopy; Conversion to Open Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group laparoscopic surgery: Participants undergo laparoscopic gastrointestinal malignancy surgery will be included in this group. The pressure of pneumoperitoneum maintain in 10-12mmHg.
  Interventions: Device: laparoscopic surgery
- group open surgery: Participants undergo open gastrointestinal malignancy surgery will be included in this group.
  Interventions: Device: open surgery

INTERVENTIONS:
Device: laparoscopic surgery — the method of surgery is conducted by laparoscope with proper pressure of pneumoperitoneum instead of opening the abdomen.
  Groups: group laparoscopic surgery
Device: open surgery — the method of surgery is conducted by surgical instruments to open the abdomen.
  Groups: group open surgery

SUMMARY:
Deep vein thrombosis (DVT) is a common complication of surgery, which could result in pulmonary embolism (PE). PE is a serious and potentially life-threatening syndrome. The purpose of this study is to investigate the impact of laparoscopic versus open surgeries on the incidence of postoperative DVT in patients with gastrointestinal malignancy

DETAILED DESCRIPTION:
Compared with open surgery (OS), the laparoscopic surgery (LS) can conduct less invasion, less pain and decrease the rate of wound infection and probably improve the quality of life for patients. For these benefits, laparoscopic surgery was widely used for gastrointestinal surgery. DVT is a common complication of surgery. However, whether LS can reduce the incidence of postoperative DVT is unclear. So the investigators conduct a cohort study, with a sufficient sample size in a rigorous scientific overview, to investigate the impact of laparoscopic versus open surgeries on the incidence of postoperative DVT in patients with gastrointestinal malignancy.

This study was approved by the institutional review board of the First Affiliated Hospital of Chongqing Medical University. The protocol design is in accordance with Consolidated Standards of Reporting Trials (CONSORT) statements.

This study is designed as a cohort study to investigate the incidence of postoperative DVT in patients undergoing gastrointestinal malignancy laparoscopic surgery (group LS) and open surgery (group OS).

Participants in group LS will receive laparoscopic gastrointestinal malignancy surgery.

Participants in group OS will receive open gastrointestinal malignancy surgery. All participants will receive unified post-operative analgesia and the prophylaxis of infection and thromboembolism.

The primary outcome of this study is the incidence of DVT after laparoscopic and open gastrointestinal malignancy surgery within 7 days postoperatively.

The secondary outcomes of this study including: concentration of plasma D - dimer 2, time to first flatus and mobility, incidence of lung infection and infection of incision within 7 days postoperatively, lengths of hospital stay .

This study will be conducted under the supervision of an independent auditor. Every week, the auditor checked the data of the participants the day after the survey was conducted. Assessment of pain intensity and prognostic outcomes must be confirmed by the auditor in sampled population. When there is disagreement between surgeon and anesthesiologists in evaluating the prognosis of patients, the auditor must solve this disagreement by discussion with both evaluators. Data were double-entered by two statisticians with limitation of access and locked during statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosed with gastrointestinal malignancy
2. aged from 18 to 75 years old
3. woman or man
4. classification of American Society of Anesthesiologists is I to III

Exclusion Criteria:

1. patients with rectal tumor need to resect anus
2. tumor distant metastasis
3. patients with palliative surgery
4. diagnosed with DVT pre-operation
5. body mass index ≤18 or ≥30
6. coagulation dysfunction
7. cerebral hemorrhage history pre-operation
8. hepatorenal dysfunction
9. being pregnant
10. mental disorder
11. patients with peritonitis or uncontrolled general infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants will be selected from the department of gastrointestinal surgery in the first affiliated hospital of chongqing medical university
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-06 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of DVT | within 7 days postoperatively
  DVT will be measured by color Doppler ultrasonography

SECONDARY OUTCOMES:
concentration of plasma D - dimer 2 | 1,3,5,7 days postoperatively
  concentration of plasma D - dimer 2 is measured by professional machine from the patients' blood
time to basic recovery | within 7 days postoperatively
  time to first flatus and mobility
incidence of lung infection | within 7 days postoperatively
  lung infection is diagnosed by X-ray ,lab examination and clinical symptoms
incidence of incision infection | within 7 days postoperatively
  incision infection is diagnosed by lab examination and clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, MD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Michota F. Venous thromboembolism: epidemiology, characteristics, and consequences. Clin Cornerstone. 2005;7(4):8-15. doi: 10.1016/s1098-3597(05)80098-5. PMID 16758647
- [Background] Nguyen NT, Owings JT, Gosselin R, Pevec WC, Lee SJ, Goldman C, Wolfe BM. Systemic coagulation and fibrinolysis after laparoscopic and open gastric bypass. Arch Surg. 2001 Aug;136(8):909-16. doi: 10.1001/archsurg.136.8.909. PMID 11485526
- [Background] Nguyen NT, Wolfe BM. The physiologic effects of pneumoperitoneum in the morbidly obese. Ann Surg. 2005 Feb;241(2):219-26. doi: 10.1097/01.sla.0000151791.93571.70. PMID 15650630
- [Background] Patel MI, Hardman DT, Nicholls D, Fisher CM, Appleberg M. The incidence of deep venous thrombosis after laparoscopic cholecystectomy. Med J Aust. 1996 Jun 3;164(11):652-4, 656. PMID 8657026
- [Background] Lord RV, Ling JJ, Hugh TB, Coleman MJ, Doust BD, Nivison-Smith I. Incidence of deep vein thrombosis after laparoscopic vs minilaparotomy cholecystectomy. Arch Surg. 1998 Sep;133(9):967-73. doi: 10.1001/archsurg.133.9.967. PMID 9749849
- [Background] Brown JA, Garlitz C, Gomella LG, McGinnis DE, Diamond SM, Strup SE. Perioperative morbidity of laparoscopic radical prostatectomy compared with open radical retropubic prostatectomy. Urol Oncol. 2004 Mar-Apr;22(2):102-6. doi: 10.1016/S1078-1439(03)00101-7. PMID 15082005
- [Background] O'Shea RT, Cook JR, Seman EI. Total laparoscopic hysterectomy: a new option for removal of the large myomatous uterus. Aust N Z J Obstet Gynaecol. 2002 Aug;42(3):282-4. doi: 10.1111/j.0004-8666.2002.00282.x. PMID 12230064
- [Background] Geerts WH, Heit JA, Clagett GP, Pineo GF, Colwell CW, Anderson FA Jr, Wheeler HB. Prevention of venous thromboembolism. Chest. 2001 Jan;119(1 Suppl):132S-175S. doi: 10.1378/chest.119.1_suppl.132s. No abstract available. PMID 11157647
- [Background] Federman DG, Kirsner RS. An update on hypercoagulable disorders. Arch Intern Med. 2001 Apr 23;161(8):1051-6. doi: 10.1001/archinte.161.8.1051. PMID 11322838
- [Background] Silver D, Vouyouka A. The caput medusae of hypercoagulability. J Vasc Surg. 2000 Feb;31(2):396-405. doi: 10.1016/s0741-5214(00)90170-8. PMID 10664508
- [Background] Wilson YG, Allen PE, Skidmore R, Baker AR. Influence of compression stockings on lower-limb venous haemodynamics during laparoscopic cholecystectomy. Br J Surg. 1994 Jun;81(6):841-4. doi: 10.1002/bjs.1800810616. PMID 8044597
- [Background] Christen Y, Reymond MA, Vogel JJ, Klopfenstein CE, Morel P, Bounameaux H. Hemodynamic effects of intermittent pneumatic compression of the lower limbs during laparoscopic cholecystectomy. Am J Surg. 1995 Oct;170(4):395-8. doi: 10.1016/s0002-9610(99)80311-0. PMID 7573736
- [Background] Ebner H, Lindemayr H. [Leg ulcer and allergic eczematous contact dermatitis incidence of contact allergies induced by topical therapy (author's transl)]. Wien Klin Wochenschr. 1977 Mar 18;89(6):185-8. German. PMID 848026
- [Background] Ido K, Suzuki T, Kimura K, Taniguchi Y, Kawamoto C, Isoda N, Nagamine N, Ioka T, Kumagai M, Hirayama Y. Lower-extremity venous stasis during laparoscopic cholecystectomy as assessed using color Doppler ultrasound. Surg Endosc. 1995 Mar;9(3):310-3. doi: 10.1007/BF00187775. PMID 7597605
- [Background] Caprini JA, Arcelus JI, Laubach M, Size G, Hoffman KN, Coats RW 2nd, Blattner S. Postoperative hypercoagulability and deep-vein thrombosis after laparoscopic cholecystectomy. Surg Endosc. 1995 Mar;9(3):304-9. doi: 10.1007/BF00187774. PMID 7597604
- [Background] Dexter SP, Griffith JP, Grant PJ, McMahon MJ. Activation of coagulation and fibrinolysis in open and laparoscopic cholecystectomy. Surg Endosc. 1996 Nov;10(11):1069-74. doi: 10.1007/s004649900242. PMID 8881054
- [Background] Filtenborg Tvedskov T, Rasmussen MS, Wille-Jorgensen P. Survey of the use of thromboprophylaxis in laparoscopic surgery in Denmark. Br J Surg. 2001 Oct;88(10):1413-6. doi: 10.1046/j.0007-1323.2001.01856.x. PMID 11578302
- [Background] Huang A, Barber N, Northeast A. Deep vein thrombosis prophylaxis protocol--needs active enforcement. Ann R Coll Surg Engl. 2000 Jan;82(1):69-70. PMID 10700773
- [Background] Schaepkens Van Riempst JT, Van Hee RH, Weyler JJ. Deep venous thrombosis after laparoscopic cholecystectomy and prevention with nadroparin. Surg Endosc. 2002 Jan;16(1):184-7. doi: 10.1007/s004640090048. Epub 2001 Oct 5. PMID 11961636
- [Background] Prevention of venous thrombosis and pulmonary embolism. NIH Consensus Development. JAMA. 1986 Aug 8;256(6):744-9. No abstract available. PMID 3723773
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271